CLINICAL TRIAL: NCT04313920
Title: Postprandial Gastric Emptying and Glycemic Response to a Pre-Operative Carbohydrate Drink in Adults With Pre-diabetes and Type II Diabetes Mellitus
Brief Title: Study of a Carbohydrate Drink in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL48
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Glycemic Response
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Supplement (Experimental): Ready to drink liquid
  Interventions: Other: Nutritional Supplement

INTERVENTIONS:
Other: Nutritional Supplement — 50 g Carbohydrate

SUMMARY:
The objective of this study is to determine the postprandial glycemic response and rates of gastric emptying in healthy subjects and those with pre-diabetes and type 2 diabetes following oral ingestion of carbohydrate.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form and provided Health Insurance Portability and Accountability Act (HIPAA) authorization
* Subject is healthy or has pre-diabetes or type 2 diabetes
* Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum
* Subject's BMI is > 18.5 kg/m2 and ≤ 40.0 kg/m2
* If subject is on a chronic medication, the dosage has been constant
* Subject states willingness to follow protocol

Exclusion Criteria:

* Subject uses exogenous insulin or Glucagon-like peptide-1 (GLP-1) receptor agonists for glucose control
* Subject has type 1 diabetes
* Subject has a history of diabetic ketoacidosis
* Subject has current infection; has had in-patient surgery, or corticosteroid treatment or antibiotics
* Subject has an active malignancy
* Subject has had a significant cardiovascular event ≤ six months or history of congestive heart failure
* Subject has end-stage organ failure or is status post organ transplant.
* Subject has a history of renal disease
* Subject has current hepatic disease
* Subject has a history of severe gastroparesis
* Subject has a chronic, contagious, infectious disease
* Subject has taken/is currently taking any herbals, dietary supplements, or medications that could profoundly affect blood glucose
* Subject has clotting or bleeding disorders
* Subject is known to be allergic or intolerant to any ingredient found in the study products
* Subject is a participant in another study that has not been approved as a concomitant study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose Concentration | Baseline 0 to 240 Minutes
  Area under the curve

SECONDARY OUTCOMES:
Serum Insulin Concentration | Baseline 0 to 240 Minutes
  Area under the curve
Nutritional Product Assessment | Immediately following product consumption
  Subject completed questionnaire with 2 product liking questions using 7-9 point Likert scale
Subjective Appetitive Ratings | Baseline 0 to 240 Minutes
  Subject completed 4 visual analog scale statements scaled from Not at All to Extremely
Gastric Emptying | Baseline 0 to 180 Minutes
  Rate of gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Cassady, PhD, RDN, LD, Study Chair — Abbott Nutrition
Locations (3):
- United States (3):
  - Health Awareness, Inc., Jupiter, Florida
  - Biofortis, Addison, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No